CLINICAL TRIAL: NCT05011214
Title: Comparison of Sedation by Esketamine and Sevoflurane for Short Ophthalmological Procedure in Children
Brief Title: Comparison of Sedation by Esketamine and Sevoflurane
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: esketamine
Record Dates: First submitted 2021-08-07; First posted 2021-08-18 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2021-08

CONDITIONS: Sevoflurane
Keywords: esketamine; sevoflurane; sedation
MeSH Terms: interventions — Sevoflurane; Esketamine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group S (Active Comparator): patients were anesthetized by face mask with 5 vol% sevoflurane with total 5 L/min-1 fresh gas flow. Anaesthesia was maintained by continuously using 3-4% sevoflurane.
  Interventions: Drug: Sevoflurane
- group E (Experimental): patients received 0.5mg/kg IV esketamine at first, after surgical field disinfection, another 0.25mg/kg IV esketamine was administered. Then 1mg/kg propofol was administered every 5 minutes after intubation.
  Interventions: Drug: Esketamine

INTERVENTIONS:
Drug: Sevoflurane — All patients received 0.01 mg/kg atropine and 1ug/kg dexmedetomidine iv as premedication.5% sevoflurane(FIO2=100%, 3L·min-1) was used to induce anaesthesia by mask inhalation and 3-4 % sevoflurane (adjusted according to the depth of the anaesthesia,FIO2=100%, 2L·min-1) was maintained
  Other Names: Sevoflurane Inhalation Solution
  Arms: group S
Drug: Esketamine — All patients received 0.1 mg/kg atropine and 1ug/kg dexmedetomidine iv as premedication.0.5mg·kg-1 esketamine was administered by vein in one minute, and 0.25mg·kg-1 esketamine was given at the beginning of the surgery.
  Other Names: s(+)ketamine
  Arms: group E

SUMMARY:
Pediatric diseases，including congenital cataract,，corneal injury，corneal ulcer, usually need suture removal and ophthalmic examination after Surgery for several days. Unfortunately, it remains a great challenge to achieve successful sedation due to children's noncooperation. Sevoflurane is one of the most often used anesthesia agents to provide deep sedation. Although sevoflurane has been used for pediatric anesthesia with successful keep spontaneous breathing without intubation, it should be noted that sevoflurane often results in air pollution under the open airway background and postoperative agitation.

Esketamine is the S (+) isomer of ketamine, which produces a dissociated state with minimal risk of airway compromise or apnea. It has enhanced analgesic potency and faster elimination compared to ketamine. However, it may also cause delirium during the recovery time. Based on these experiences on ketamine, we compared the effectiveness of esketamine and sevoflurane for short ophthalmological procedure in pediatric patients.

DETAILED DESCRIPTION:
Pediatric diseases，including congenital cataract,，corneal injury，corneal ulcer, usually need suture removal and ophthalmic examination after Surgery for several days. Unfortunately, it remains a great challenge to achieve successful sedation to avoid body movement and keep perfect eye position due to children's noncooperation. Thus, appropriate sedative agents therefore need to be administrated to perform this minor surgery. Sevoflurane is used frequently inhalational anaesthetic agent to provide pediatric anaesthesia because of the nonirritant nature. It has been used for successful keeping spontaneous breathing without tracheal intubation. It should be noted that sevoflurane often results in air pollution under the open airway background and emergence agitation. High concentrations of sevoflurane may causes respiratory depression due to the decrease in tidal volume during spontaneous ventilation.

Ketamine is widely used for procedural sedation, which produces a dissociated state with minimal risk of airway compromise or apnea. Esketamine is the S (+) isomer of ketamine, It has enhanced analgesic potency and faster elimination compared to ketamine. However, it may also cause agitation during the recovery time. Based on these experiences on ketamine, we compared the effectiveness of esketamine and sevoflurane for short ophthalmological procedure in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* patient who needed suture removal and ophthalmic examination

Exclusion Criteria:

* previous coronary heart disease,hypertension, arterial aneurysm, epilepsia, intracranial mass of benign or malign nature

Ages: 3 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-20 (Estimated)

PRIMARY OUTCOMES:
eye position scale | during the surgery
  1=The inner and outer canthus line across the central cornea; 2= Inferior limbus does not exceed the inner and outer canthus line; 3= Inferior limbus exceed the inner and outer canthus line.

SECONDARY OUTCOMES:
the incidence of respiratory depression | during the surgery
  decreased tidal volume or weak chest undulation
the incidence of desaturation | during the surgery
  the incidence of oxygen saturation below 95% caused by anesthetic agents
Intraocular pressure | the time after intubation and topical anesthesia within 1 minute
  Intraocular pressure after induction
requirements for additional propofol | during the surgery
  If the target level of sedation was not achieved, an additional 0.1mg/kg propofol was injected and repeated if necessary
CPS score | scores at the time point of 1 minutes after extubation
  The Cole 5-point scale (CPS) score included five behaviors: 1=sleeping; 1=awake,calm;3=irritable, crying;4=inconsolable crying; 5=severe restlessness, disorientation.
length of stay in the post-anesthesia care unit | duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 20 mins
  the time of the length of stay in the post-anesthesia care unit
Mean blood pressure pressure | 1minutes before induction;1minutes after induction;1minutes before intubation;1minutes after intubation,3 minutes after intubation
  mean blood pressure
Heart rate | 1minutes before induction;1minutes after induction;1minutes before extubation;1minutes after extubation,3 minutes after extubation
  Heart rate
extubation time | duration from the time that patients arrived in post-anesthesia care unit to the time of extubation, average 10 mins
  extubation time

CONTACTS AND LOCATIONS:
Overall Officials: Fang Tan, Principal Investigator — Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University
Locations (1):
- Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Green SM, Roback MG, Kennedy RM, Krauss B. Clinical practice guideline for emergency department ketamine dissociative sedation: 2011 update. Ann Emerg Med. 2011 May;57(5):449-61. doi: 10.1016/j.annemergmed.2010.11.030. Epub 2011 Jan 21. PMID 21256625
- [Result] Cao Q, Lin Y, Xie Z, Shen W, Chen Y, Gan X, Liu Y. Comparison of sedation by intranasal dexmedetomidine and oral chloral hydrate for pediatric ophthalmic examination. Paediatr Anaesth. 2017 Jun;27(6):629-636. doi: 10.1111/pan.13148. Epub 2017 Apr 17. PMID 28414899
- [Result] Krishnappa S, Kundra P. Optimal anaesthetic depth for LMA insertion. Indian J Anaesth. 2011 Sep;55(5):504-7. doi: 10.4103/0019-5049.89887. PMID 22174469